CLINICAL TRIAL: NCT03498365
Title: Effects of the Use of Multi Criterion Decision Analysis (MCDA) on Decision Quality in an Online Delphi
Acronym: Delphi-MCDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ThinkWell (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Amy Price, Principal Investigator, ThinkWell
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PLOT-D MCDA
Record Dates: First submitted 2018-04-01; First posted 2018-04-13 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Behavioral Changes
Keywords: decision analysis; decision support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online MCDA (Experimental)
  Interventions: Behavioral: MCDA
- Online Delphi (Active Comparator)
  Interventions: Behavioral: Delphi

INTERVENTIONS:
Behavioral: MCDA — Experimental decision support
  Arms: Online MCDA
Behavioral: Delphi — Standard support
  Arms: Online Delphi

SUMMARY:
To examine the effects of using decision support tools during the online Delphi process.

DETAILED DESCRIPTION:
The purpose of this exploratory work is to develop improved methods for building a protocol for a participatory randomized controlled trial. An online Delphi will be combined with an embedded trial testing the effectiveness of a decision support tool. This method provides for consensus building and collaborative problem-solving which is informed, and participatory. The online Delphi offers involvement and confidentiality thus sidestepping the complications of power imbalances and undue influence as respondents contribute anonymously.

The embedded trial was considered after the building of a database of existing online trials and conducting a descriptive analysis" Creating a database of Internet-based clinical trials to support a public-led research programme: A descriptive analysis, followed by the completion of a systematic overview of systematic overviews, "Patient and Public Involvement in Clinical Trials Design: An Overview of Systematic Reviews" and followed this with an analysis of "Self-Management Open Online Trials in Health"(In review). The results included a lack of standardization, insufficient guidance for implementation and significant research reporting weaknesses. Decision-making support tools may improve decision quality.

This embedded trial will be implemented in an online Delphi to come to the consensus about what declarations and methods to include when building a participatory online trials protocol.

ELIGIBILITY:
Inclusion Criteria:

Protocol lab online trialsl Delphi (PLOT-D) Participant

Exclusion Criteria:

* None if meets inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
My Decision Quality (MDQ) | Up to 20 weeks or study completion
  MDQ is a patient reported outcome measure that combines a set of importance weights for multiple criteria (options, effect, importance, chance, trust, support ,control and commitment) with performance ratings for each option on these criteria and calculates the overall score as the expected value of these components.

OTHER OUTCOMES:
Time to consensus | Up to 20 weeks or study completion
  Aggregated group time to reach consensus

CONTACTS AND LOCATIONS:
Overall Officials: Amy I Price, PhD, Principal Investigator — University of Oxford; Mike J Clarke, DPhil, Principal Investigator — Queen's University, Belfast; Mette Kjer Kaltoft, PhD, Study Director — Syddansk Universitet; Jack Dowie, PhD, Study Director — The London School of Hygiene & Tropical Medicine
Locations (1):
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data is not available due to data protection rules. De-identified aggregated data may be available by contacting the Principal Investigator
Supporting Information: Study Protocol, ICF
Time Frame: following publication
Access Criteria: contact PI

REFERENCES:
- [Background] Price A, Albarqouni L, Kirkpatrick J, Clarke M, Liew SM, Roberts N, Burls A. Patient and public involvement in the design of clinical trials: An overview of systematic reviews. J Eval Clin Pract. 2018 Feb;24(1):240-253. doi: 10.1111/jep.12805. Epub 2017 Oct 27. PMID 29076631
- [Background] Brice A, Price A, Burls A. Creating a database of internet-based clinical trials to support a public-led research programme: A descriptive analysis. Digit Health. 2015 Nov 20;1:2055207615617854. doi: 10.1177/2055207615617854. eCollection 2015 Jan-Dec. PMID 29942546
- [Background] Dowie J, Kjer Kaltoft M, Salkeld G, Cunich M. Towards generic online multicriteria decision support in patient-centred health care. Health Expect. 2015 Oct;18(5):689-702. doi: 10.1111/hex.12111. Epub 2013 Aug 2. PMID 23910715
- [Background] Kaltoft MK, Dowie J, Turner R, et al. Decisional equipoise is not decisional conflict: avoiding the false clarity bias in the evaluation of decision aids and Shared Decision Making processes. F1000Research 2015;4. doi:10.7490/F1000RESEARCH.1110671.1
- [Background] Kaltoft M, Cunich M, Salkeld G, Dowie J. Assessing decision quality in patient-centred care requires a preference-sensitive measure. J Health Serv Res Policy. 2014 Apr;19(2):110-7. doi: 10.1177/1355819613511076. Epub 2013 Dec 12. PMID 24335587